CLINICAL TRIAL: NCT06076213
Title: Efficacy and Safety of Artesunate-amodiaquine and Artemether-lumefantrine in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in the Democratic Republic of the Congo: a Randomized Controlled Trial (TES2022)
Brief Title: Test Efficacy Study on the Recommended Antimalarial Drugs in the Democratic Republic of the Congo
Acronym: TES2022
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Global Fund (Other)
Responsible Party: Principal Investigator, Prof. Gauthier Mesia Kahunu, Professor, Ministry of Public Health, Democratic Republic of the Congo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASAQ-AL 2022
Record Dates: First submitted 2023-09-24; First posted 2023-10-10 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: Uncomplicated malaria; Plasmodium falciparum; Artemisinin-based Combination Treatment; Artemether-lumefantrine; Artesunate-amodiaquine
MeSH Terms: conditions — Malaria, Falciparum | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 in two treatment arms: artesunate-amodiaquine and artemether-lumefantrine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artesunate-amodiaquine (Experimental): tablets of ASAQ Winthrop®
  Interventions: Drug: Artesunate-amodiaquine
- Artemether-lumefantrine (Experimental): tablets of Coartem Dispersible®
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artesunate-amodiaquine — Tablets
  Other Names: ASAQ Winthrop®
  Arms: Artesunate-amodiaquine
Drug: Artemether-lumefantrine — Tablets
  Other Names: Coartem Dispersible®
  Arms: Artemether-lumefantrine

SUMMARY:
Malaria remains a public health concern, despite efforts that are invested in the disease control. The Democratic Republic of the Congo (DRC) is one of the most affected countries in Sub Saharan Africa. Artemisinin-based combination treatments (ACTs) are recommended for the treatment of uncomplicated malaria. However, reported cases of mutations that confer to Plasmodium falciparum resistance to artemisinin (the main component of ACTs) constitute a threat to malaria control, particularly in Sub Saharan Africa. Therefore, the recommendation of the World Health Organization to conduct regularly test efficacy studies in endemic countries is paramount.

The purpose of this trial is to assess efficacy and safety of artesunate-amodiaquine (ASAQ Winthrop®) and artemether-lumefantrine (Coartem Dispersible®) at day 28 for the treatment of uncomplicated Plasmodium falciparum malaria in eight surveillance sites around DRC.

DETAILED DESCRIPTION:
This is a phase IV, randomized, open label, 2-arm trial. It will be performed in eight malaria sentinel sites around DRC. Children aged 6 to 59 months with confirmed Plasmodium falciparum uncomplicated malaria will be enrolled after informed consent granted by a parent or guardian. They will be randomized to receive either artesunate-amodiaquine or artemether lumefrantrine during 3 days (directly observed treatment) and then followed up until day 28. At each visit, clinical examination (including collection of safety data) will be done and malaria testing as well. Dried blood spots will also be prepared whenever microscopy is performed, in order to assess resistance markers and perform the genotyping of the parasite for PCR-adjusted efficacy. Hemoglobin level will be measured on the recruitment day and then every two weeks until day 28.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 to 59 months
* monoinfection with Plasmodium falciparum with asexual parasite count of 2,000 to 200,000/µL
* axillary temperature ≥ 37.5 °C
* ability to swallow oral medication
* ability and willingness to comply with the protocol for the duration of the study and to comply with the study visit schedule;
* informed consent from a parent or a guardian
* living within the study catchment area
* absence of severe manutrition
* absence of infectious diseases that can be responsible of fever
* absence of allergy to the study drugs

Exclusion Criteria:

* presence of general danger signs or signs of severe falciparum malaria according to the definitions of WHO;
* body weight < 5kg
* hemoglobin level < 5g/ dL or hematocrit < 15%
* presence of severe malnutrition
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* malaria treatment within 2 days prior to recruitment
* history of hypersensitivity reactions or contraindications to any of the medicines being tested or used as alternative treatment;
* body weight below 5 kg

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1260 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
PCR adjusted efficacy | day 28
  Absence of fever and negative blood smear during the follow-up until day 28 or new infection occurred during the follow-up.

SECONDARY OUTCOMES:
Proportion of adverse events and serious adverse events | day 28
  Number of adverse events and serious adverse events that every participant will experience
Prevalence of HRP2 deletion | Baseline
  Proportion of positive samples that fail to be detected by malaria rapid diagnostic tests due to the deletion of the related antigen
Prevalence of resistance markers at baseline | Baseline
  Proportion of samples containing different markers of resistance to different antimalarial drugs
Quantification of Lumefantrine | day 7
  Level of lumefantrine in the blood of children who will be randomized to the Artemether-lumefantrine arm

CONTACTS AND LOCATIONS:
Locations (7):
- Democratic Republic of the Congo (7):
  - Centre de santé de Coopération, Kimpese, Bas-Congo Province
  - Centre de santé Lupidi 1, Kapolowe, Haut-Katanga
  - Centres de santé de Mikalayi et Matamba, Kazumba, Kasai-Central
  - Centre de Santé de Vanga, Vanga, Kwilu
  - Centre de santé de Kalima, Kalima, Maniema Province
  - Centres de santé Umoja et Foyer social, Kabondo, Tshopo
  - Centre de santé Boende 2 Nsele, Boende, Tshuapa